CLINICAL TRIAL: NCT06795243
Title: Efficacy of Physical Therapy Treatment in Endometriosis and Its Relationship to Adherence Rates.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Manuel Rebollo Salas, Principal investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SICEIA 2024-146
Record Dates: First submitted 2025-01-11; First posted 2025-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis; Endometriosis Related Pain; Endometriosis, Pain; Endometriosis-related Pain; Pain; Pain Intensity Assessment; Pain Management; Pain, Chronic Disease; Pain Score; Therapeutic Exercise; Exercise Adherence; Adherence, Treatment; Treatment Adherence and Compliance; Quality of Life
Keywords: Endometriosis; Endometriosis Related Pain; Endometriosis, Pain; Pain; Pain Intensity Assessment; Pain Management; Pain, chronic disease; pain score; therapeutic exercise; exercise adherence; Adherence, Treatment; Treatment Adherence and Compliance; Quality of life
MeSH Terms: conditions — Endometriosis; Pain; Agnosia; Chronic Disease; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Application of a multimodal physical therapy program based on pain education and therapeutic exercise. Sixteen sessions will be carried out. The sessions will be carried out with a frequency of two days a week. Subjects will receive 6 PAIN NEUROSCIENCE EDUCATION (PNE), and 8 weeks (2 times/ week) of therapeutic exercise.
  Interventions: Procedure: PAIN NEUROSCIENCE EDUCATION AND THERAPEUTIC EXERCISE PROGRAM
- Control Group (Active Comparator): Usual Care. Application of standard medical treatment. In Spain, the treatment provided is mainly pharmacological, adjusted to the symptomatic profile of theses patients.
  Interventions: Procedure: USUAL CARE

INTERVENTIONS:
Procedure: PAIN NEUROSCIENCE EDUCATION AND THERAPEUTIC EXERCISE PROGRAM — PAIN NEUROSCIENCE EDUCATION
  1. Introduction to the knowledge of pain in the XXI century. Pain as an alarm system.
  Types of pain. Differences between acute and chronic pain. 3. Chronic pain. Concepts of kinesiophobia, catastrophism and fear avoidance, self-determination and neuroplasticity.
  4. Main pain management tools based on scientific evidence. 5. . Transtheoretical model of change. Adherence to treatment, importance as a determinant in health.
  6. Messages for home. Strategies of active coping in the maintenance stage.
  THERAPEUTIC EXERCISE PROGRAM 10-min warm-up. Joint mobility exercises with dual task or gamification. 30-min main part. Sequence of balance work between strength and body flexibility dosed according to the specific needs of each participant.
  10-min cool down including breathing exercises and motor imagery. Home exercise program: walking (150 minutes in total, 3 days alternating with the face-to-face sessions).
  Arms: Experimental Group
Procedure: USUAL CARE — The treatment provided is mainly pharmacological, adjusted to the symptomatic profile of theses patients.
  Conventional medical care is based on hormonal, pharmacological and/or surgical treatment and is carried out on an individualized basis depending on the severity of the disease and the patient's needs, especially in matters of desire to become pregnant. Surgical treatment is carried out when pharmacological therapy (hormonal or anti-inflammatory) is ineffective or involves adverse events.
  Arms: Control Group

SUMMARY:
The main objective of this study is to know if the application of both therapies, neuroscience pain education plus therapeutic exercise will modify pain, catastrophizing and quality of life in endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic and inflammatory gynecological condition characterized by the growth of endometrial- like tissue within and outside the pelvic cavity (uterus).

With current means and diagnostic systems, a prevalence of 10% is estimated, although the evidence warns that with the improvement of early diagnosis, these figures will be much higher in the future. One of the main problems with endometriosis is the late diagnosis, which takes an average of seven years. Added to this is the fact that until a definitive diagnosis, patients live in the adolescent stage with symptoms (around 50% with severe pelvic pain) that cause disability and changes in activity and participation in daily life.

At the social level, endometriosis patients are known to have limitations in academic and work activities, as well as in social participation. All of this causes high economic costs.

Chronic pelvic pain can cause the phenomenon of central nervous system sensitization in which pain processing is altered. Pain catastrophizing significantly affects pain disability and vice versa in endometriosis.

Conventional medical care is based on hormonal, pharmacological, and / or surgical treatment and is carried out on an individualized basis depending on the severity of the treatment and the patient's needs.

The multidisciplinary approach to endometriosis has gained relevance in recent decades and has been considered by leaders in the clinical and research sectors. Within the multidisciplinary team, physiotherapy has gained relevance in recent decades.

The multimodal approach of physiotherapy is the one that the Clinical Practice Guidelines and national and international documents demand with greater relevance. Therapeutic exercise based on the work of the abdominal stabilizing musculature and motor control appears to be effective in the treatment of nonspecific low back pain and in endometriosis-related pain. But there is no 'gold standard' in terms of dosage, considering the individualization of treatments.

In the biopsychosocial care paradigm, and specifically in the approach to pathologies with primary chronic pain, patients tend to be motivated and accompanied toward self-determination to achieve adherence to treatment through health education strategies, adequate information, and personalized and goal-oriented multimodal treatment.

However, today, nonadherence is positioned as a global problem, which is growing as the burden of chronicity of pathologies increases, influencing health outcomes and long-term healthcare costs.

Due to symptomatology especially related to chronic pain in endometriosis and in the context of the biopsychosocial paradigm demanded by the scientific community, the investigators consider pertinent the study of catastrophization and its relationship with quality of life and, therefore, disability, and an intervention that addresses in a multimodal way the physiotherapy treatment for endometriosis.

It is recognized that physiotherapeutic interventions based on therapeutic exercise programs, both individual and group, are most effective when tailored to the needs of everyone. Part of this customization should focus on the barriers that each patient recognizes to treatment adherence.

For this reason, the investigators found that studies that support further research to increase the basic understanding of the factors that act as a barrier to adherence in physical therapy treatments could facilitate the development of strategies to overcome nonadherence. And if the investigators follow international recommendations, these systems should address adherence and compliance to treatment from a multidimensional perspective.

Therefore, the investigators believe that measuring compliance and adherence to treatment in this way in patients with endometriosis would allow to know whether adherence to the proposed exercise programs in the target population and their effectiveness are really related or not to the adherence rates to treatment as suggested in recent publications.

In view of the above, this project aims to examine the relationship between the efficacy of physical therapy treatment in patients diagnosed with endometriosis measured in clinical and quality of life terms with short-term compliance and short- and medium-term adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (over 18 years of age) diagnosed with endometriosis.
* Women with the capacity to carry out a therapeutic program based on muscular exercise.
* Women with the capacity to understand the requirements of the study.

Exclusion Criteria:

* Women undergoing fertility and/or assisted reproduction treatment.
* Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Self-report Pain magnitude | At the start of the study (at baseline, 0 week), 1 month and 2 months after the start of the intervention (4 and 8 weeks), 1 month from the last session (12th week), 3 months from the last session (20th week) and 6 months from the last session (32th week
  Magnitude of chronic pain: Chronic pain grading scale. Likert-type scale with 8 items that are evaluated between 0 and 10 for items 2, 3, 4, 6, 7 and 8. Item 1 collects the number of days with pain in the last six months. Item 5 rates the impediment to the performance of usual tasks in the last three months, and can be evaluated between none and 90. The higher the score, the greater the chronic pain involvement. If the score is zero, the patient will be rated as having no pain. Chronic pain will be of low interference with grade I (low intensity) or grade II (high intensity) or of high interference with grade III (moderately limiting) or grade IV (severely limiting). Persistence will be graded as non-persistent or persistent pain.
Treatment Compliance | From enrollment to the end of treatment at 8 weeks
  Self-report of the person responsible for managing attendance at the group sessions in the experimental group. Participants who attend 80% or more of the sessions will be considered compliant.
Treatment adherence (Maintenance of the therapeutic exercise program at home ) | From the end of the intervention at 8 weeks (starting at week 9) to the end of treatment at 32 weeks
  Adherence to treatment (experimental group), measured by visual analogue scale (VAS) included in the patient diary, in terms of:
  Maintenance of treatment at home: number of days that the proposed exercise is performed (100% being 3 times a week). Each patient will complete the VAS scale weekly. Participants with a score equal to or greater than 80 points out of 100 on the VAS scale will be considered to have high adherence.
Changes from Self-report pain catastrophizing | At the start of the study (at baseline, 0 week), 1 month and 2 months after the start of the intervention (4 and 8 weeks), 1 month from the last session (12th week), 3 months from the last session (20th week) and 6 months from the last session (32th week
  Catastrophizing thoughts in the face of pain: Pain Catastrophizing Scale (PCS). Pain catastrophizing is a construct that is related to a negative and exaggerated orientation towards painful stimuli. The scale, validated in Spanish, is a list of 13 statements that describe different thoughts and feelings that may be related to pain in the dimensions of rumination, magnification and hopelessness. The person indicates the degree to which he/she has such thoughts or feelings by rating them between 0 (not at all) and 4 (all the time). The theoretical range of the instrument is between 13 and 62, with higher values indicating a higher index of catastrophizing.
Change from Self-report specific quality of life | At the start of the study (at baseline, 0 week), 1 month and 2 months after the start of the intervention (4 and 8 weeks), 1 month from the last session (12th week), 3 months from the last session (20th week) and 6 months from the last session (32th week
  Specific quality of life: Endometriosis Health Profile (EHP-30+23) questionnaire Spanish version. The questionnaire is composed of two parts. Part 1 with 30 itmens and part 2 divided into five subscales: pain, control and helplessness, emotional well-being, social support and self-image. For part 1 and each subscale a total score is created as a percentage of the maximum possible score. 0 is considered the best possible health status and 100 the worst.
Changes in self-reported general quality of life | At the start of the study (at baseline, 0 week), 1 month and 2 months after the start of the intervention (4 and 8 weeks), 1 month from the last session (12th week), 3 months from the last session (20th week) and 6 months from the last session (32th week
  Overall Quality of Life: EUROQOL-5 Dimensions- 3 Levels (EQ-5D-3L). It is a standardized instrument that measures health outcomes and is applicable to a wide range of diseases and treatments. It provides a simple descriptive profile and a single index of health status. The EQ-5D-3L covers 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is assessed in 3 categories (no problems; moderate problems; extreme problems). The assessment consists of measuring each of the 5 domains in one of the 3 categories. In this work we use, as in our reference study, the validated Spanish version of the EQ-5D-3L in its current version for the adult population. EQ-5D © 2025 EuroQol Research Foundation.

SECONDARY OUTCOMES:
Exercise-related adverse events | At the start of the study (at baseline, 0 week), 1 month and 2 months after the start of the intervention (4 and 8 weeks), 1 month from the last session (12th week), 3 months from the last session (20th week) and 6 months from the last session (32th week
  Possible occurrence of pain, frequency of flares and fatigue, measured qualitatively in narrative text through patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen-María Suárez-Serrano, Study Chair — Departamento de Fisioterapia. Facultad de Enfermería, Fisioterapia y Podología de la Universidad de Sevilla.; José-Jesús Jiménez-Rejano, Study Director — Departamento de Fisioterapia. Facultad de Enfermería, Fisioterapia y Podología de la Universidad de Sevilla.; Manuel Rebollo-Salas, Study Director — Departamento de Fisioterapia. Facultad de Enfermería, Fisioterapia y Podología de la Universidad de Sevilla.; Inmaculada Villa-del-Pino, Principal Investigator — Centro universitario San Isidoro, adscrito a Universidad Pablo de Olavide, Sevilla.
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
  The data to be provided will refer to all the variables of the study: independent, dependent and control variables.
  Dependent (Catastrophic thoughts about pain, magnitude of chronic pain, general quality of life, specific quality of life, adverse events related to exercise ( pain, frequency of flares and fatigue), adherence and compliance to treatment Control variables:
  * Age (years).
  * Height: measured in centimeters.
  * Weight: measured in kilograms.
  * BMI: (kg/m2).
  * Work and/or academic activity: measured according to whether the person works, studies or both at the same time.
  * Academic level: measured according to whether the person has compulsory or higher education.
  * Stage of pathology: measured in stages according to the American Society for Reproductive Medicine.
  All this will be carried out preserving the confidentiality of the data of the study participants according to the rules of the Ethics Committee of the University of Seville.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available in the repository of the University of Seville once the research has been completed and the research report has been written.

REFERENCES:
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Bordeleau M, Vincenot M, Lefevre S, Duport A, Seggio L, Breton T, Lelard T, Serra E, Roussel N, Neves JFD, Leonard G. Treatments for kinesiophobia in people with chronic pain: A scoping review. Front Behav Neurosci. 2022 Sep 20;16:933483. doi: 10.3389/fnbeh.2022.933483. eCollection 2022. PMID 36204486
- [Background] Hamacher D, Hamacher D, Schega L. A cognitive dual task affects gait variability in patients suffering from chronic low back pain. Exp Brain Res. 2014 Nov;232(11):3509-13. doi: 10.1007/s00221-014-4039-1. Epub 2014 Jul 25. PMID 25059910
- [Background] Fernandez-Rodriguez R, Alvarez-Bueno C, Cavero-Redondo I, Torres-Costoso A, Pozuelo-Carrascosa DP, Reina-Gutierrez S, Pascual-Morena C, Martinez-Vizcaino V. Best Exercise Options for Reducing Pain and Disability in Adults With Chronic Low Back Pain: Pilates, Strength, Core-Based, and Mind-Body. A Network Meta-analysis. J Orthop Sports Phys Ther. 2022 Aug;52(8):505-521. doi: 10.2519/jospt.2022.10671. Epub 2022 Jun 19. PMID 35722759
- [Background] Galan-Martin MA, Montero-Cuadrado F, Lluch-Girbes E, Coca-Lopez MC, Mayo-Iscar A, Cuesta-Vargas A. Pain Neuroscience Education and Physical Therapeutic Exercise for Patients with Chronic Spinal Pain in Spanish Physiotherapy Primary Care: A Pragmatic Randomized Controlled Trial. J Clin Med. 2020 Apr 22;9(4):1201. doi: 10.3390/jcm9041201. PMID 32331323
- [Background] Mari-Alexandre J, Garcia-Oms J, Agababyan C, Belda-Montesinos R, Royo-Bolea S, Varo-Gomez B, Diaz-Sierra C, Gonzalez-Canto E, Gilabert-Estelles J. Toward an improved assessment of quality of life in endometriosis: evaluation of the Spanish version of the Endometriosis Health Profile 30. J Psychosom Obstet Gynaecol. 2022 Sep;43(3):251-257. doi: 10.1080/0167482X.2020.1795827. Epub 2020 Jul 31. PMID 32735156
- [Background] Jones GL, Budds K, Taylor F, Musson D, Raymer J, Churchman D, Kennedy SH, Jenkinson C. A systematic review to determine use of the Endometriosis Health Profiles to measure quality of life outcomes in women with endometriosis. Hum Reprod Update. 2024 Mar 1;30(2):186-214. doi: 10.1093/humupd/dmad029. PMID 38007607
- [Background] Ferrer-Pena R, Gil-Martinez A, Pardo-Montero J, Jimenez-Penick V, Gallego-Izquierdo T, La Touche R. Adaptation and validation of the Spanish version of the graded chronic pain scale. Reumatol Clin. 2016 May-Jun;12(3):130-8. doi: 10.1016/j.reuma.2015.07.004. Epub 2015 Aug 19. English, Spanish. PMID 26298083
- [Background] Wheeler CHB, Williams ACC, Morley SJ. Meta-analysis of the psychometric properties of the Pain Catastrophizing Scale and associations with participant characteristics. Pain. 2019 Sep;160(9):1946-1953. doi: 10.1097/j.pain.0000000000001494. PMID 30694929
- [Background] Xu Y, Deng Z, Fei F, Zhou S. An overview and comprehensive analysis of interdisciplinary clinical research in endometriosis based on trial registry. iScience. 2024 Feb 20;27(3):109298. doi: 10.1016/j.isci.2024.109298. eCollection 2024 Mar 15. PMID 38455973
- [Background] Tennfjord MK, Gabrielsen R, Tellum T. Effect of physical activity and exercise on endometriosis-associated symptoms: a systematic review. BMC Womens Health. 2021 Oct 9;21(1):355. doi: 10.1186/s12905-021-01500-4. PMID 34627209
- [Background] Tourny C, Zouita A, El Kababi S, Feuillet L, Saeidi A, Laher I, Weiss K, Knechtle B, Zouhal H. Endometriosis and physical activity: A narrative review. Int J Gynaecol Obstet. 2023 Dec;163(3):747-756. doi: 10.1002/ijgo.14898. Epub 2023 Jun 22. PMID 37345574
- [Background] McLean SM, Burton M, Bradley L, Littlewood C. Interventions for enhancing adherence with physiotherapy: a systematic review. Man Ther. 2010 Dec;15(6):514-21. doi: 10.1016/j.math.2010.05.012. Epub 2010 Jul 14. PMID 20630793
- [Background] Jack K, McLean SM, Moffett JK, Gardiner E. Barriers to treatment adherence in physiotherapy outpatient clinics: a systematic review. Man Ther. 2010 Jun;15(3):220-8. doi: 10.1016/j.math.2009.12.004. Epub 2010 Feb 16. PMID 20163979
- [Background] Nagpal TS, Mottola MF, Barakat R, Prapavessis H. Adherence is a key factor for interpreting the results of exercise interventions. Physiotherapy. 2021 Dec;113:8-11. doi: 10.1016/j.physio.2021.05.010. Epub 2021 Sep 21. PMID 34555674
- [Background] Rubi-Carnacea F, Masbernat-Almenara M, Climent-Sanz C, Soler-Gonzalez J, Garcia-Escudero M, Martinez-Navarro O, Valenzuela-Pascual F. Effectiveness of an exercise intervention based on preactivation of the abdominal transverse muscle in patients with chronic nonspecific low back pain in primary care: a randomized control trial. BMC Prim Care. 2023 Sep 6;24(1):180. doi: 10.1186/s12875-023-02140-3. PMID 37674205
- [Background] Wojcik M, Szczepaniak R, Placek K. Physiotherapy Management in Endometriosis. Int J Environ Res Public Health. 2022 Dec 2;19(23):16148. doi: 10.3390/ijerph192316148. PMID 36498220
- [Background] Artacho-Cordon F, Salinas-Asensio MDM, Galiano-Castillo N, Ocon-Hernandez O, Peinado FM, Mundo-Lopez A, Lozano-Lozano M, Alvarez-Salvago F, Arroyo-Morales M, Fernandez-Lao C, Cantarero-Villanueva I. Effect of a Multimodal Supervised Therapeutic Exercise Program on Quality of Life, Pain, and Lumbopelvic Impairments in Women With Endometriosis Unresponsive to Conventional Therapy: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Nov;104(11):1785-1795. doi: 10.1016/j.apmr.2023.06.020. Epub 2023 Jul 17. PMID 37467936
- [Background] Abril-Coello R, Correyero-Leon M, Ceballos-Laita L, Jimenez-Barrio S. Benefits of physical therapy in improving quality of life and pain associated with endometriosis: A systematic review and meta-analysis. Int J Gynaecol Obstet. 2023 Jul;162(1):233-243. doi: 10.1002/ijgo.14645. Epub 2023 Jan 17. PMID 36571475
- [Background] Goncalves AV, Barros NF, Bahamondes L. The Practice of Hatha Yoga for the Treatment of Pain Associated with Endometriosis. J Altern Complement Med. 2017 Jan;23(1):45-52. doi: 10.1089/acm.2015.0343. Epub 2016 Nov 21. PMID 27869485
- [Background] Mardon AK, Leake HB, Hayles C, Henry ML, Neumann PB, Moseley GL, Chalmers KJ. The Efficacy of Self-Management Strategies for Females with Endometriosis: a Systematic Review. Reprod Sci. 2023 Feb;30(2):390-407. doi: 10.1007/s43032-022-00952-9. Epub 2022 Apr 29. PMID 35488093
- [Background] Aredo JV, Heyrana KJ, Karp BI, Shah JP, Stratton P. Relating Chronic Pelvic Pain and Endometriosis to Signs of Sensitization and Myofascial Pain and Dysfunction. Semin Reprod Med. 2017 Jan;35(1):88-97. doi: 10.1055/s-0036-1597123. Epub 2017 Jan 3. PMID 28049214
- [Background] Levang SL, Pukall CF. An Investigation of Associations between Pain Catastrophizing and Pain Disability in a Diverse Sample of Persons with Endometriosis. J Obstet Gynaecol Can. 2024 Apr;46(4):102340. doi: 10.1016/j.jogc.2023.102340. Epub 2024 Jan 1. PMID 38171483
- [Background] Hemmert R, Schliep KC, Willis S, Peterson CM, Louis GB, Allen-Brady K, Simonsen SE, Stanford JB, Byun J, Smith KR. Modifiable life style factors and risk for incident endometriosis. Paediatr Perinat Epidemiol. 2019 Jan;33(1):19-25. doi: 10.1111/ppe.12516. Epub 2018 Oct 11. PMID 30307628
- [Background] Salinas-Asensio MDM, Ocon-Hernandez O, Mundo-Lopez A, Fernandez-Lao C, Peinado FM, Padilla-Vinuesa C, Alvarez-Salvago F, Postigo-Martin P, Lozano-Lozano M, Lara-Ramos A, Arroyo-Morales M, Cantarero-Villanueva I, Artacho-Cordon F. 'Physio-EndEA' Study: A Randomized, Parallel-Group Controlled Trial to Evaluate the Effect of a Supervised and Adapted Therapeutic Exercise Program to Improve Quality of Life in Symptomatic Women Diagnosed with Endometriosis. Int J Environ Res Public Health. 2022 Feb 2;19(3):1738. doi: 10.3390/ijerph19031738. PMID 35162761
- [Background] Armour M, Sinclair J, Chalmers KJ, Smith CA. Self-management strategies amongst Australian women with endometriosis: a national online survey. BMC Complement Altern Med. 2019 Jan 15;19(1):17. doi: 10.1186/s12906-019-2431-x. PMID 30646891
- [Background] Horne AW, Missmer SA. Pathophysiology, diagnosis, and management of endometriosis. BMJ. 2022 Nov 14;379:e070750. doi: 10.1136/bmj-2022-070750. PMID 36375827
- [Background] Parsons BA, Baranowski AP, Berghmans B, Borovicka J, Cottrell AM, Dinis-Oliveira P, Elneil S, Hughes J, Messelink BEJ, de C Williams AC, Abreu-Mendes P, Zumstein V, Engeler DS. Management of chronic primary pelvic pain syndromes. BJU Int. 2022 May;129(5):572-581. doi: 10.1111/bju.15609. Epub 2021 Oct 27. PMID 34617386
- [Background] Lara-Ramos A, Alvarez-Salvago F, Fernandez-Lao C, Galiano-Castillo N, Ocon-Hernandez O, Mazheika M, Salinas-Asensio MM, Mundo-Lopez A, Arroyo-Morales M, Cantarero-Villanueva I, Artacho-Cordon F. Widespread Pain Hypersensitivity and Lumbopelvic Impairments in Women Diagnosed with Endometriosis. Pain Med. 2021 Sep 8;22(9):1970-1981. doi: 10.1093/pm/pnaa463. PMID 33675228
- [Background] Biggs WS, Carey ET, McIntyre JM. Limited evidence guides empiric Tx of female chronic pelvic pain. J Fam Pract. 2018 Mar;67(3):E1-E9. PMID 29509818
- See also: Related Info — https://www.consejo-fisioterapia.org/adjuntos/publicaciones/publicacion_2.pdf
- See also: Related Info — https://www.aetsa.org/download/publicaciones/Endometriosis_DEF.pdf
- See also: Related Info — https://www.sspa.juntadeandalucia.es/servicioandaluzdesalud/sites/default/files/sincfiles/wsas-media-mediafile_sasdocumento/2019/guia_endometriosis_2018.pdf
- See also: Related Info — https://www.sanidad.gob.es/organizacion/sns/planCalidadSNS/pdf/equidad/ENDOMETRIOSIS.pdf
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK11822/